CLINICAL TRIAL: NCT03525899
Title: Macular Hole After Diabetic Vitrectomy
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201709039RINB
Record Dates: First submitted 2018-04-08; First posted 2018-05-16 (Actual); Last update posted 2018-05-16 (Actual); Status verified 2017-10

CONDITIONS: Proliferative Diabetic Retinopathy; Macular Holes
MeSH Terms: conditions — Retinal Perforations

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MH after diabetic pars plana vitrectomy: Recruited patients included, the persistent MH group, who had MH before the primary DV, and the newly-developed MH group, who developed MH after a successful primary DV
  Interventions: Procedure: Pars plana vitrectomy

INTERVENTIONS:
Procedure: Pars plana vitrectomy — Pars plana vitrectomy combined with Internal limiting membrane peeling, inverted internal limiting membrane flap insertion into the macular hole, or lens anterior or posterior capsular flap insertion into the macular hole

SUMMARY:
To present the clinical characteristics and rational treatment of macular hole (MH) after the diabetic vitrectomy (DV) in patients with proliferative diabetic retinopathy (PDR).

DETAILED DESCRIPTION:
All patients had received initial vitrectomy to treat complications of PDR. Recruited patients were divided to two groups: the persistent MH group, who had MH before the primary DV (group 1); and the newly-developed MH group, who developed MH after a successful primary DV (group 2). The patients' demographic data, records of ophthalmological examinations, and surgical procedures were collected, including best-corrected visual acuity before and after each operation, fundus changes, as well as MH repairing techniques. The extent of fibrovascular proliferation(FVP) was separated into four grades based on the severity of vitreoretinal adhesion : multiple-point adhesions with or without one site plaque-like broad adhesion (grade 1), broad adhesions in more than one but fewer than three sites, located posterior to the equator (grade 2), broad adhesions in more than three sites, located posterior to the equator or extending beyond the equator within one quadrant (grade 3), and broad adhesions extending beyond the equator for more than one quadrant (grade 4). The extent of retinal detachment (RD) was classified into "within the arcade" or "beyond the arcade". The macular structure was evaluated by optical coherence tomography (OCT). All patients had a follow-up duration of more than three months after the final surgical procedures.

Three different surgical techniques were used to treat MH: standard internal limiting membrane (ILM) peeling, inverted ILM flap insertion into the MH, and lens anterior or posterior capsular flap insertion into the MH. The indication(s) for each technique were:

standard ILM peeling was performed if no ILM peeling had been done in the previous surgery, and the MH size was less than 500um in an attached retina; inverted ILM flap insertion was performed if no ILM peeling had been done in the previous surgery, with a detached retina; lens anterior capsule flap insertion was performed if cataract surgery was performed in the same setting with no ILM tissue available; lens posterior capsule flap insertion was performed in a pseudophakic eye with no ILM tissue available. Only descriptive statistics was obtained.

ELIGIBILITY:
Inclusion Criteria:

* Proliferative diabetic retinopathy patients presenting with macular hole after primary diabetic vitrectomy
* The persistent MH group after surgery, who had MH before the primary DV
* Newly-developed MH group, who developed MH after a successful primary diabetic retinopathy

Exclusion Criteria:

* Patients with peripheral breaks
* Patients with macular hole before surgery, which closed after primary diabetic retinopathy
* Missing clinical data

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from January 2010 to May 2017 treated by a single surgeon (Y.C.M) at National Taiwan University Hospital were retrospectively reviewed.
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
Time to macular hole closure | OCT was performed monthly after operation, until MH closure was achieved, up yo 1 year
  Evaluation by optical coherence tomography

SECONDARY OUTCOMES:
Best corrected visual acuity | One month after operation, and then the visual acuity was checked every six months. Up to 3.5 years.
  Landolt C chart

CONTACTS AND LOCATIONS:
Overall Officials: Chung-May Yang, MD, Study Director — National Taiwan University Hospital
Locations (1):
- Department of Ophthalmology, National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Yeh PT, Cheng CK, Chen MS, Yang CH, Yang CM. Macular hole in proliferative diabetic retinopathy with fibrovascular proliferation. Retina. 2009 Mar;29(3):355-61. doi: 10.1097/IAE.0b013e31818c3251. PMID 18997639
- [Background] Chen SN, Yang CM. LENS CAPSULAR FLAP TRANSPLANTATION IN THE MANAGEMENT OF REFRACTORY MACULAR HOLE FROM MULTIPLE ETIOLOGIES. Retina. 2016 Jan;36(1):163-70. doi: 10.1097/IAE.0000000000000674. PMID 26200509
- [Background] Ghoraba H. Types of macular holes encountered during diabetic vitrectomy. Retina. 2002 Apr;22(2):176-82. doi: 10.1097/00006982-200204000-00007. PMID 11927850